CLINICAL TRIAL: NCT05315596
Title: Longitudinal Assessment of Pain-related Patient-reported Outcomes in the Sub-acute Phase After Surgery: a Registry Study From PAIN OUT
Brief Title: Longitudinal Assessment of Pain-Related Patient-Reported Outcomes After Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán (Unknown); Centro Medico Nacional Siglo XXI IMSS (Other); Hospital de Traumatología y Ortopedia Lomas Verdes (Unknown); Hospital Angeles Puebla (Unknown); Hospital General de Chihuahua - Dr. Salvador Zubirán Anchondo (Other Government); Hospital Angeles Lomas (Other); Hospital San Javier Guadalajara (Unknown); Hospital Aranda de La Parra (Leon Guanajuato) (Unknown); Fundación Clínica Médica Sur (Other); Instituto Nacional de Cancerologia de Mexico (Other); Hospital General Dr. Ruben Leñero (Other); Hospital Central "Dr. Ignacio Morones Prieto" (Other); Hospital General Regional Número 2 Dr. Guillermo Fajardo Ortiz (Unknown); Instituto Nacional de Enfermedades Respiratorias (Other Government); Hospital Central Militar (Other Government)
Responsible Party: Principal Investigator, Ruth Zaslansky, PAIN OUT - scientific director, Jena University Hospital
Other Study IDs: JenaUH_pain
Record Dates: First submitted 2022-02-23; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Adult; Pain Measurement; Functional Status; Pain Management; Neuralgia; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Little is known about pain-related outcomes experienced by patients in the first few weeks after surgery, once they are discharged from hospital.

This study aims to characterize pain, pain-related interference, and early neuropathic pain in the sub-acute phase after surgery.

DETAILED DESCRIPTION:
A high proportion of patients experience moderate to severe pain after surgery. However, most of the knowledge about this comes from studies where patients are evaluated in the hours and up until the first postoperative day. Alternatively, patients are assessed several months (eg 3 or later) after surgery, to evaluate the development of chronic pain related to surgery (CPSP) and most patients do not develop CPSP.

This study aims to learn how patients recover concerning pain and function once they return home after surgery. How long is it before they can resume their daily activities and to do so in comfort? Do they take treatment for pain? Do they have pain restricted to the surgical incision or it is more widespread? There is little knowledge as to whether there are signs of nerve injury in the days close to surgery. This type of pain might lead to chronic pain in later stages.

Patients will be assessed at three time points: the first day after surgery, the 7th day after surgery, and 1 month.

The information we obtain will offer healthcare providers, from multiple hospitals, information about the care they provide to their patients for pain while patients are still in hospital and insights as to how the care might be improved, once they are discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Adult
2. On the first post-operative day and back on the ward for at least 6 hours
3. Gives consent for assessment at 3-time points

Exclusion Criteria:

1. The patient is unable to communicate
2. The patient is cognitively impaired
3. The patient is asleep
4. The patient is too ill or in too much pain and does not wish to be interviewed
5. The patient does not wish to fill in the outcomes questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients after surgery
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in pain interference scores between postoperative day 7 (POD7) and 1 month after surgery (POM1). | 7th day after surgery (POD7) and 1 Month (M1) after surgery
  We will assess whether pain-related functional impairment on postoperative day 7 is associated with functional pain-related impairment 1 month after surgery. Functional pain impairment will be assessed using the BPI short-form questionnaire and calculated as a Pain Interference Total Score (PITS) from the 7 interference questions in the BPI. Patients will be allocated to groups of no (PITS=0)/mild-(PITS=1-2)/ moderate /(PITS=2-5) and severe interference (PITS>5). Mean scores of the 2 domains within the functional items, physical interference (general activity, walking ability, and work) and effective interference (mood, enjoyment of life, and relations with other persons) will also be calculated. Sleep will addressed separately as it does not improve psychometric properties of the BPI interference scale. This methodology has been used in another PAIN OUT study, evaluating function at 6 months after surgery (Stamer et al, Pain. 2019 Aug;160(8):1856-1865).
The number of patients with high pain interference on the 7th day after surgery (POD7). | Day 7 after surgery
  Number of patients with high pain interference at postoperative day 7 (POD7, BPI-PITS >5).

SECONDARY OUTCOMES:
Differences in pain severity (BPI-PSVS, pain severity scale) between postoperative day 7 and 1 month after surgery (POM1). | Day 7 after surgery and Month 1 after surgery
  We will use the pain severity variables in the BPI to assess pain on postoperative day 7 compared to Month 1 after surgery.
The differences in pain interference (BPI-PITS) between surgical disciplines on postoperative day 7. | Day 7 after surgery
  This will be a cohort of patients undergoing surgeries from different disciplines. We anticipate that median pain interference scores will not differ between the disciplines.
The differences in pain interference (BPI-PITS) between surgical disciplines at month 1 after surgery. | 1 Month after surgery
  This will be a cohort of patients undergoing surgeries from different disciplines. We anticipate that median pain interference scores will not differ between the disciplines.
The difference in the number of patients with signs of neuropathy on postoperative day 7 between the surgical disciplines. | Day 7 after surgery
  The difference in the number of patients with signs of neuropathy on postoperative day 7 (DN2 score ≥ 3/7) between the surgical disciplines.
  Neuropathy will be screened for using the 'Douleur Neuropathique en 2 Questions' (DN2) . Neuropathy is indicated for a score of >3/7 items in the questionnaire (Beloeil et al Early postoperative neuropathic pain assessed by the DN4 score predicts an increased risk of persistent postsurgical neuropathic pain. Eur J Anesthesiology 2017;34:652-7).
The difference in the number of patients with signs of neuropathy at 1 month after surgery (POM1) between the surgical disciplines. | 1 Month after surgery
  The difference in the number of patients with signs of neuropathy at POM1 (DN2 score ≥ 3/7) between the surgical disciplines.
Differences in pain interference scores between patients with vs without signs of neuropathy on postoperative day 7 | Day 7 after surgery
  Differences in pain interference (BPI-PITS) between patients with vs. without signs of neuropathy (DN2 score ≥ 3/7) on postoperative day 7.
Differences in pain interference (BPI-PITS) between patients with vs. without signs of neuropathy (DN2 score ≥ 3/7) at POM1. | 1 Month after surgery
  Differences in pain interference (BPI-PITS) between patients with vs. without signs of neuropathy (DN2 score ≥ 3/7) at POM1.
Differences in pain severity between patients with vs without signs of neuropathy at POM1 | 1 Month after surgery
  Differences in pain severity (BPI-PSVS) between patients with vs. without signs of neuropathy (DN2 score ≥ 3/7) at POM1.
Assess the difference in the number of patients taking analgesics o POD7 vs POD1. | Day 7 after surgery and 1 Month after surgery
  The difference in the number of patients taking analgesics between postoperative day 7 and POM1. Patients will be asked if they are taking an analgesic at both time points.

OTHER OUTCOMES:
Exploratory regression analysis for improving understanding of pain interference on day 7 after surgery | First postoperative day and postoperative day 7
  Exploratory regression analysis for pain interference on postoperative day 7 (BPI-PITS, dependent variable), demographic variables, perioperative treatment variables and patient-reported outcomes (International Pain Out Questionnaire) from the first post-operative day (POD1).
Exploratory regression analysis for improving understanding of pain intensity on postoperative day 7. | First postoperative day and postoperative day 7
  Exploratory regression analysis for pain intensity on postoperative day 7 (BPI-PSVS, dependent variable). Independent variables will include demographic variables, perioperative treatment variables and patient-reported outcomes obtained on the first postoperative day (POD1)
Exploratory regression analysis for improving understanding of pain intensity at POM1 | First postoperative day and 1 month after surgery
  Exploratory regression analysis for pain intensity at POM1 (BPI-PSVS, dependent variable). Independent variables will include: demographic variables, perioperative treatment variables and patient reported outcomes (International Pain Out Questionnaire) from the first postoperative day (POD1).

CONTACTS AND LOCATIONS:
Overall Officials: Ana L Garduño López, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Vicotor M Acosta-Nava, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Ruth Zaslansky, DSc, Principal Investigator — Jena University Hospital
Locations (16):
- Jena University Hospital, Jena, Germany
- Mexico (15):
  - Hospital General de Chihuahua Salvador Zubirán Anchondo, El Bajo, Chihuahua
  - Hospital Aranda de La Parra (Leon Guanajuato), León, Guanajuato
  - Hospital Central Militar, Mexico City, Mexico City
  - Hospital San Javier Guadalajara, Guadalajara
  - Centro Nacional SIGLO XXI (IMSS), Mexico City
  - Hospital Angeles Interlomas CDMX, Mexico City
  - Hospital de traumatologia y Ortopedia Lomas Verdes (IMSS), Mexico City
  - Hospital fundación Medica Sur, Mexico City
  - Hospital General de Villacoapa (IMSS), Mexico City
  - Hospital Ruben Leñero, Mexico City
  - Instituto Nacional de Cancerología, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias Cosio Villegas (INER), Mexico City
  - Hospital Angeles Puebla, Puebla City
  - Hospital Central Morones Prieto San Luis Potosi, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: Undecided
Data collected by each hospital belongs to them.

REFERENCES:
- See also: Website of PAIN OUT, a perioperative pain registry and research network — http://www.pain-out.eu